CLINICAL TRIAL: NCT05916469
Title: Heavy Menstrual Bleeding Progestin Treatment in Bleeding Disorders Study
Acronym: HMB-BD
Status: Recruiting | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: University of Washington (Other); NIH National Heart, Lung, and Blood Institute (Unknown)
Responsible Party: Principal Investigator, Maureen Baldwin, Associate Professor of Ob/Gyn, Oregon Health and Science University
Other Study IDs: LNG-IUD BD Study
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Heavy Menstrual Bleeding; Bleeding Disorder; Von Willebrand Diseases
MeSH Terms: conditions — Menorrhagia; Hemostatic Disorders; von Willebrand Diseases | interventions — Levonorgestrel; Norethindrone Acetate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Bleeding disorder using LNG-IUD: Adolescents and young adults ages 10-24 with diagnosed bleeding disorder planning use of LNG-IUD.
  Interventions: Drug: Levonorgestrel Intrauterine System
- Non-bleeding disorder using LNG-IUD: Adolescents and young adults ages 10-24 without diagnosed bleeding disorder planning use of LNG-IUD.
  Interventions: Drug: Levonorgestrel Intrauterine System
- Bleeding disorder using NETA: Adolescents and young adults ages 10-24 with diagnosed bleeding disorder planning use of NETA.
  Interventions: Drug: Norethindrone Acetate

INTERVENTIONS:
Drug: Levonorgestrel Intrauterine System — 52 mg levonorgestrel intrauterine system
  Other Names: Mirena; Liletta
  Groups: Bleeding disorder using LNG-IUD; Non-bleeding disorder using LNG-IUD
Drug: Norethindrone Acetate — norethindrone acetate 5 mg daily
  Other Names: Aygestin
  Groups: Bleeding disorder using NETA

SUMMARY:
The goal of this multicenter prospective observational study and registry of U.S. adolescents and young adults with heritable bleeding disorders is to determine the bleeding outcomes, satisfaction, hemostatic parameter changes, and patient reported quality of life after 6 months of use of either of two commonly used hormonal treatments for menstrual suppression - levonorgestrel intrauterine device (LNG-IUD) and norethindrone acetate (NETA). Under this application the study will compare the two treatments and compare outcomes after LNG-IUD treatment results to a control group without a bleeding disorder, with the goal of determining the benefits and expected outcomes of these treatment options for this population.

DETAILED DESCRIPTION:
Heavy menstrual bleeding (HMB) is common among adolescents and young adults with an inherited bleeding disorder (BD) and negatively impacts health-related quality of life and physical and mental health status. Effective treatment options are available that decrease bleeding and improve quality of life, but were not studied in those with BD, so investigators do not know if there is similar effectiveness in this condition. The impact of treatment on diagnostic testing for BD or on improvement of iron deficiency is also not known. Given these gaps in knowledge, the primary objective of the Heavy Menstrual Bleeding Progestin Treatment in Bleeding Disorders Study is to conduct a multicenter prospective observational cohort study and registry, enrolling adolescents and young adults with heavy menstrual bleeding cared for at collaborating interdisciplinary menstrual clinic sites nationally who are choosing to start use of either of two commonly used progestin menstrual treatment options: levonorgestrel-releasing intrauterine system (LNG-IUD) or oral norethindrone acetate 5 mg daily (NETA) (N=300). In Aim 1, the study will compare outcomes related to (a) bleeding management, (b) quality of life, and (c) repletion of iron storage levels after six months of treatment with either option in those with a diagnosed inherited bleeding disorder. The primary outcome will be treatment success with a Pictorial Blood Loss Assessment Chart (PBAC) score <50 points by six months. Secondary objectives to assess bleeding management will include need for adjuvant management, change in PBAC from baseline to 6 months, and self-reported treatment success. Quality of life outcomes will include change in validated scales to assess health-related quality of life which are specific to adolescents and young adults in the setting of heavy menstrual bleeding. The study will compare ferritin levels at six months compared to baseline to determine the relative amount of benefit obtained from either treatment option. In Aim 2, the study will compare outcomes after LNG-IUD in those with and without a bleeding disorder, assessing rates of expulsion and method continuation between the two groups in addition to the outcomes assessed for Aim 1. Aim 3 will improve our understanding of the impact of physiological stress on BD diagnostic studies by comparing change in hemostatic parameters before and after successful treatment in those with HMB without a previously diagnosed bleeding disorder. This study will demonstrate the relative benefits of menstrual suppression treatment options for adolescents and young adults with heavy menstrual bleeding and inherited bleeding disorders, will provide population-specific estimates for expected benefit that can be used in treatment counseling, and will highlight the impact of treatment status on diagnostic test results.

ELIGIBILITY:
Inclusion Criteria:

* Post-menarcheal
* Ages 10-24
* Decision to initiate a trial of progestin therapy with either LNG-IUD or NETA
* Able to provide assent and written informed consent by one parent (ages <18) or written informed consent (age 18+)
* Must meet trial criteria for heavy menstrual bleeding
* Must meet trial criteria for a bleeding disorder or have minimum workup to rule out bleeding disorder

Exclusion Criteria:

* Pregnant or seeking pregnancy

Ages: 10 Years to 24 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents and young adults ages 10-24 with and without a heritable bleeding disorder who receive medical care for heavy menstrual bleeding at a participating U.S. clinical site. All clinical sites participate in a national consortium of interdisciplinary hematology-gynecology clinics.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-09-24 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Treatment success rate | 6 months
  Proportion with pictorial blood loss assessment score <50 points

SECONDARY OUTCOMES:
Median Pictorial Blood Assessment Chart (PBAC) score | 6 months
  Group median of pictorial blood loss assessment score. PBAC scores start at 0 to represent no bleeding with higher PBAC scores representing heavy menstrual bleeding. There is no maximum PBAC score.
Patient-reported treatment success rate | 6 months
  Proportion with patient-reported treatment success. Treatment success will be measured with Yes or No bivariate response.
Change in Adolescent Menstrual Bleeding Questionnaire (aMBQ) score | Baseline to 6 months
  Group median of individual change in adolescent menstrual bleeding questionnaire score. aMBQ scores can range from 0 to 77 with higher scores representing worse health-related quality of life.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS-25 or PROMIS-29) scores | Baseline to 6 months
  Group median of individual change in patient-reported outcomes measurement information system score after treatment. PROMIS-25 and PROMIS-29 scores are measured on a standardized scale of T-scores with a score of 50 representing the population average and higher scores representing worse outcomes. Participants who will be age 18 or older at six months after treatment initiation will be administered the PROMIS-25 adult version and age <18 will be administered the PROMIS-29 pediatric version.
Change in serum ferritin after treatment | Baseline to 6 months
  Group median of individual change in ferritin
Change in von Willebrand Factor (VWF) levels | Baseline to 6 months
  Group median of individual change in von Willebrand Factor levels

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Baldwin, MD MPH, Principal Investigator — Oregon Health and Science University; Allison Wheeler, Principal Investigator — University of Washington
Locations (9):
- United States (9):
  - Stanford, Palo Alto, California
  - Colorado Anschutz Medical Campus, Aurora, Colorado
  - Emory, Atlanta, Georgia
  - University of Michigan Medicine, Ann Arbor, Michigan
  - Children's Mercy, Kansas City, Missouri
  - Oregon Health & Science University, Portland, Oregon
  - Penn State Health, Hershey, Pennsylvania
  - University of Washington, Seattle, Washington
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
This study will collect clinical, laboratory, and survey data from participants ages 10-24 at multiple academic clinical sites. Participant-level clinical data will be preserved through deposition of the data in a controlled access public repository. We will make our scientific data as widely and freely available as possible while safeguarding the privacy of participants (de-identified prior to repository submission) and protecting confidential and proprietary data.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Scientific data will be shared as soon as possible following study participant completion. Scientific data included in published manuscripts will be available at the time of publication; all other generated scientific data will be shared no later than the end of the award. The study data will be stored in the repository indefinitely, for at least 5 years.
Access Criteria: The study datasets will be collected with the following informed consent: The dataset can only be used for studying health, medical, or biomedical conditions and does not include the study of population origins or ancestry. We will also require all individuals requesting data to enter into a data sharing agreement that: 1) acknowledges the data will be stripped of identifying markers and identification; 2) acknowledges that these data will only be used for research purposes; and 3) requests investigators to reference the seminal publication describing data collection. The dataset can only be used for studying health, medical or biomedical conditions and does not include the study of population origins or ancestry. The requesting institution's IRB or equivalent body must approve the requested use.